CLINICAL TRIAL: NCT04858581
Title: Prospective Clinical and Virological Analysis of Healthcare Workers Diagnosed Positive for Covid-19.
Acronym: Pro-Co-HPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-A02720-39
Record Dates: First submitted 2021-04-15; First posted 2021-04-26 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Serologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthcare workers who had a diagnosis confirmed by a nasopharyngeal RT-PCR test with SARS-CoV-2 (Other): Survey, RT-PCR test and blood test.
  Interventions: Diagnostic Test: Virological and serological tests

INTERVENTIONS:
Diagnostic Test: Virological and serological tests — Survey, RT-PCR test and blood test

SUMMARY:
Coronavirus disease 2019 (COVID-19) is an acute infection of the respiratory tract that emerged in late 2019.

In several studies, the cardinal signs of COVID-19 associated fever, cough, sputum and dyspnea occurring in the first days of infection. In addition, myalgia was frequent (14.9-32.3%) and digestive signs which may be inaugural were also reported, such as diarrhea (3.8-5%) and nausea/vomiting (4-5%).

An increase in medical consultations for anosmia and ageusia without nasal obstruction has also been reported in the context of the COVID-19.

Mild or non-existent symptoms, but also serious forms leading to death or a long stay in intensive care, within a few months, the multiple clinical signs of SARS-CoV-2 infection were identified. But, beyond the acute symptoms, doctors and patients are discovering a whole range of disorders occurring more distantly, in hospitalized patients or not. In this context of an emerging viral infection such as SARS-CoV-2, many unknowns are still present such as the duration of symptoms or post-infectious sequelae in patients.

DETAILED DESCRIPTION:
The scientific and medical world is mobilizing to accelerate the production of knowledge on this virus, on the disease it causes as well as the means of curing and preventing it. But no one yet knows how much it can cause immunological changes in the body. For some specialists, this virus is even much more than a viral infection and causes a general disruption of the immune system.

Faced with the COVID-19 pandemic, healthcare workers are a particularly exposed.

The main objective of this research is to assess the presence of symptoms attributed to COVID-19 at least 6 months after infection confirmed by RT-PCR test of healthcare workers.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers over 18 years of age
* Healthcare workers who had a diagnosis confirmed by a nasopharyngeal RT-PCR test with SARS-CoV-2
* Healthcare workers with signed consent

Exclusion Criteria:

* Protected healthcare workers
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Description of symptoms attributed to COVID-19 at 6 months. | 6 months after COVID-19 infection
  The primary outcome is the description of symptoms attributed to COVID-19 at least 6 months after infection confirmed by RT-PCR test.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Gagnard, Principal Investigator — Hôpital privé d'Antony
Locations (1):
- Hopital privé d'Antony, Paris, France

IPD SHARING:
Plan to Share IPD: No